CLINICAL TRIAL: NCT03805919
Title: Natural History Study of Men at High Genetic Risk for Prostate Cancer
Brief Title: Men at High Genetic Risk for Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190040; 19-C-0040
Record Dates: First submitted 2019-01-15; First posted 2019-01-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12-02

CONDITIONS: Prostatic Neoplasms
Keywords: BRCA 1; BRCA 2; MMR genes; Lynch Syndrome; Natural History
MeSH Terms: conditions — Prostatic Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with germline pathogenic or likely pathogenic variants in prostate cancer-related risk genes

SUMMARY:
Background:

Research studies have shown that genetic changes and family history may increase a man s risk for prostate cancer. Researchers want to follow the prostate health of men who have specific genetic changes associated with prostate cancer to help them learn more about which men are at higher risk for prostate cancer.

Objectives:

To study men with specific genetic changes and determine who is at higher risk for getting prostate cancer. To study if certain genetic changes and family history can be used to help prevent or treat prostate cancer.

Eligibility:

Males between ages 30-75 who have one or more specific genetic changes but without prostate cancer.

Design:

* This study does not perform genetic testing. All participants must have documented genetic changes and able to provide a copy of the report.
* Before enrollment, participants will provide a copy of documented genetic changes and go through a telephone interview to determine eligibility for the study.
* On enrollment, participants will have medical and family history review, medication review, physical exam, blood collection for clinical and research testing, and MRI (magnetic resonance imaging) of the prostate.
* Every year, participants will repeat the physical exam, medical history, family history, medication review, routine blood tests, including PSA and testosterone.
* Every 2 years, participants will repeat all the above plus prostate MRI and blood tests for research.
* If, at any time, the physical exam, blood tests or MRI are abnormal, participants may be asked to do a biopsy.
* If the biopsy results in prostate cancer, participants will be given counseling on next steps, general treatment recommendations, and then followed with a phone call each year.
* Participants may ask to speak with a genetic counselor.

DETAILED DESCRIPTION:
Background:

Prostate cancer is the most common malignancy and the second leading cause of cancer-related deaths in American men.

Prostate cancer has substantial inherited predisposition and certain genetic variants that are associated with an increased risk of prostate cancer.

An evolving approach to prostate cancer screening is to target populations at risk of developing prostate cancer based on their genetic predisposition.

Objective:

To follow the natural history of men with known germline variants or likely pathogenic variants in genes that put them at risk for developing prostate cancer.

Eligibility:

Males between ages 30-75 years old.

Documented germline pathogenic or likely pathogenic variants in prostate cancer-related risk gene: BRCA 1 and 2, DNA Mismatch Repair (MMR) genes associated with Lynch syndrome (MLH1, MSH2, MSH6, PMS2, and EPCAM), HOXB13, ATM, NBN, TP53, CHEK2, PALB2, RAD51C, RAD51D, BRIP1, or FANC (FANCA, FANCB, FANCC, FANCD2, FANCE, FANCF, FANCG, FANCI, FANCL, and FANCM).

Must be able and willing to provide informed consent.

Design:

Up to 500 subjects will be enrolled.

Participants will undergo sampling of blood for prostate-specific antigen. Based on these results and age, participants will be considered for biopsy and/or continued monitoring if feasible upon clinical discretion.

Participants will undergo a baseline MRI evaluation with follow-up scans every 2 years as clinically indicated.

Following initial evaluation, participants will be followed as clinically indicated, usually at 12 month intervals, to determine their PSA level, prostate cancer treatment (if relevant) and/or disease/survival status until death.

ELIGIBILITY:
* Inclusion Criteria:
* Males between ages 30-75 years old.
* Documented germline variant (i.e. pathogenic/likely pathogenic variant) in prostate cancer risk-related gene from a CLIA certified laboratory: BRCA1 and BRCA2, MMR genes (MLH1, MSH2, MSH6, PMS2, and EPCAM) associated with Lynch syndrome, as well as HOXB13, ATM, NBN, TP53, CHEK2, PALB2, RAD51C, RAD51D, BRIP1, or FANC (FANCA, FANCB, FANCC, FANCD2, FANCE, FANCF, FANCG, FANCI, FANCL, and FANCM).
* Prognosis of >5 years survival if affected by another cancer
* Ability of subject to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior diagnosis or treatment for prostate cancer
* Known contraindication to MRI:

  * Participants unable to fit through MRI scanner (radiologist discretion)
  * Allergy to MR contrast agent
  * Participants with pacemakers, cerebral aneurysm clips, shrapnel injury, or implantable electronic device
* Active concomitant medical or psychological illnesses that may increase the risk to the subject or inability to obtain informed consent, at the discretion of the principal investigator.

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with a documented germline variant in prostate cancer risk-related gene from a CLIA certified laboratory
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2039-01-01 (Estimated)

PRIMARY OUTCOMES:
Natural history of high genetic risk for prostate cancer | one year
  To follow the natural history of men with known germline variants or likely pathogenic variants in genes that put them at high risk for developing prostate cancer

SECONDARY OUTCOMES:
mpMRI feasibility | baseline and every two years until death or when criteria for removal from study is met
  test the feasibility and accuracy of multi parametric magnetic resonance imaging (mpMRI) for the localization and detection of local prostate cancer
role of mpMRI | baseline and every two years until death or when criteria for removal from study is met
  role of mpMRI in monitoring participants on active surveillance and as a follow up tool for monitoring local disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Fatima H Karzai, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
-All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@-In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: -Clinical data available during the study and indefinitely.@@@@@@-Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: -Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@-Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Al Olama AA, Kote-Jarai Z, Berndt SI, Conti DV, Schumacher F, Han Y, Benlloch S, Hazelett DJ, Wang Z, Saunders E, Leongamornlert D, Lindstrom S, Jugurnauth-Little S, Dadaev T, Tymrakiewicz M, Stram DO, Rand K, Wan P, Stram A, Sheng X, Pooler LC, Park K, Xia L, Tyrer J, Kolonel LN, Le Marchand L, Hoover RN, Machiela MJ, Yeager M, Burdette L, Chung CC, Hutchinson A, Yu K, Goh C, Ahmed M, Govindasami K, Guy M, Tammela TL, Auvinen A, Wahlfors T, Schleutker J, Visakorpi T, Leinonen KA, Xu J, Aly M, Donovan J, Travis RC, Key TJ, Siddiq A, Canzian F, Khaw KT, Takahashi A, Kubo M, Pharoah P, Pashayan N, Weischer M, Nordestgaard BG, Nielsen SF, Klarskov P, Roder MA, Iversen P, Thibodeau SN, McDonnell SK, Schaid DJ, Stanford JL, Kolb S, Holt S, Knudsen B, Coll AH, Gapstur SM, Diver WR, Stevens VL, Maier C, Luedeke M, Herkommer K, Rinckleb AE, Strom SS, Pettaway C, Yeboah ED, Tettey Y, Biritwum RB, Adjei AA, Tay E, Truelove A, Niwa S, Chokkalingam AP, Cannon-Albright L, Cybulski C, Wokolorczyk D, Kluzniak W, Park J, Sellers T, Lin HY, Isaacs WB, Partin AW, Brenner H, Dieffenbach AK, Stegmaier C, Chen C, Giovannucci EL, Ma J, Stampfer M, Penney KL, Mucci L, John EM, Ingles SA, Kittles RA, Murphy AB, Pandha H, Michael A, Kierzek AM, Blot W, Signorello LB, Zheng W, Albanes D, Virtamo J, Weinstein S, Nemesure B, Carpten J, Leske C, Wu SY, Hennis A, Kibel AS, Rybicki BA, Neslund-Dudas C, Hsing AW, Chu L, Goodman PJ, Klein EA, Zheng SL, Batra J, Clements J, Spurdle A, Teixeira MR, Paulo P, Maia S, Slavov C, Kaneva R, Mitev V, Witte JS, Casey G, Gillanders EM, Seminara D, Riboli E, Hamdy FC, Coetzee GA, Li Q, Freedman ML, Hunter DJ, Muir K, Gronberg H, Neal DE, Southey M, Giles GG, Severi G; Breast and Prostate Cancer Cohort Consortium (BPC3); PRACTICAL (Prostate Cancer Association Group to Investigate Cancer-Associated Alterations in the Genome) Consortium; COGS (Collaborative Oncological Gene-environment Study) Consortium; GAME-ON/ELLIPSE Consortium; Cook MB, Nakagawa H, Wiklund F, Kraft P, Chanock SJ, Henderson BE, Easton DF, Eeles RA, Haiman CA. A meta-analysis of 87,040 individuals identifies 23 new susceptibility loci for prostate cancer. Nat Genet. 2014 Oct;46(10):1103-9. doi: 10.1038/ng.3094. Epub 2014 Sep 14. PMID 25217961
- [Background] Haraldsdottir S, Hampel H, Wei L, Wu C, Frankel W, Bekaii-Saab T, de la Chapelle A, Goldberg RM. Prostate cancer incidence in males with Lynch syndrome. Genet Med. 2014 Jul;16(7):553-7. doi: 10.1038/gim.2013.193. Epub 2014 Jan 16. PMID 24434690
- [Background] Giri VN, Knudsen KE, Kelly WK, Abida W, Andriole GL, Bangma CH, Bekelman JE, Benson MC, Blanco A, Burnett A, Catalona WJ, Cooney KA, Cooperberg M, Crawford DE, Den RB, Dicker AP, Eggener S, Fleshner N, Freedman ML, Hamdy FC, Hoffman-Censits J, Hurwitz MD, Hyatt C, Isaacs WB, Kane CJ, Kantoff P, Karnes RJ, Karsh LI, Klein EA, Lin DW, Loughlin KR, Lu-Yao G, Malkowicz SB, Mann MJ, Mark JR, McCue PA, Miner MM, Morgan T, Moul JW, Myers RE, Nielsen SM, Obeid E, Pavlovich CP, Peiper SC, Penson DF, Petrylak D, Pettaway CA, Pilarski R, Pinto PA, Poage W, Raj GV, Rebbeck TR, Robson ME, Rosenberg MT, Sandler H, Sartor O, Schaeffer E, Schwartz GF, Shahin MS, Shore ND, Shuch B, Soule HR, Tomlins SA, Trabulsi EJ, Uzzo R, Vander Griend DJ, Walsh PC, Weil CJ, Wender R, Gomella LG. Role of Genetic Testing for Inherited Prostate Cancer Risk: Philadelphia Prostate Cancer Consensus Conference 2017. J Clin Oncol. 2018 Feb 1;36(4):414-424. doi: 10.1200/JCO.2017.74.1173. Epub 2017 Dec 13. PMID 29236593
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-C-0040.html